CLINICAL TRIAL: NCT01078688
Title: Evaluation of the Frequency of Limitation of Activity, Depending on Gender and Age-group, in Patients With Persistent Asthma Consulting a General Practitioner
Brief Title: Evaluation of the Frequency of Limitation of Activity in Patients With Persistent Asthma
Acronym: ASMAVIE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RFR-DUM-2009/2
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Persistent Asthma
Keywords: Limitations of activities; persistent asthma; general practitioner; frequency of limitations of activities; depending on gender and age-group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the frequency of limitation of activity, depending on gender and age-group, in patients with persistent asthma consulting a general practitioner

ELIGIBILITY:
Inclusion Criteria:

* persistent asthma receiving long-term maintenance treatment with inhaled steroids (alone or in combination with other drugs)

Exclusion Criteria:

* Patients with a diagnosis of COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First 3 consecutive patients with persistent asthma seen by general practitioner receiving long-term maintenance treatment with inhaled steroids
Sampling Method: Probability Sample
Enrollment: 1942 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To describe the frequency of limitations of activities in patients with persistent asthma depending on gender and age-group. | Last 3 months / once
To describe, depending on gender and age-group, the nature of the activities limited, the degree of limitation and the impact on the patient's daily life. | Once during only visit

SECONDARY OUTCOMES:
To describe the nature of the activities limited, the degree of limitation and the impact on the patient's daily life according to the level of asthma control | Once during only visit
To describe, depending on gender and age-group, the activities that need to be specifically investigated in routine clinical practice due to their greater impact on the patient's quality of life, and which could indicate poorly controlled asthma | Once during only visit
To describe the main characteristics and initial management for all patients of the survey | Once during only visit

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, Study Director — AstraZeneca
Locations (724):
- France (724):
  - Research Site, Abbaretz
  - Research Site, Abbeville
  - Research Site, Achenheim
  - Research Site, Achicourt
  - Research Site, Afa
  - Research Site, Aiguillon
  - Research Site, Aixe-sur-Vienne
  - Research Site, Ajaccio
  - Research Site, Albertville
  - Research Site, Albi
  - Research Site, Ambès
  - Research Site, Ambierle
  - Research Site, Andance
  - Research Site, Andernos-les-Bains
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Anizy-le-Château
  - Research Site, Annonay
  - Research Site, Arches
  - Research Site, Aregno
  - Research Site, Arles
  - Research Site, Ars
  - Research Site, Art-sur-Meurthe
  - Research Site, Asnières-sur-Seine
  - Research Site, Aubenas
  - Research Site, Aubervilliers
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Auchy-les-Mines
  - Research Site, Audincourt
  - Research Site, Audruicq
  - Research Site, Aulnat
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aurillac
  - Research Site, Autun
  - Research Site, Auxi-le-Château
  - Research Site, Avesnes-le-Sec
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Baignes Ste Radegonde
  - Research Site, Bailly
  - Research Site, Balma
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Basse-Goulaine
  - Research Site, Bassillac
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Bâgé-le-Châtel
  - Research Site, Beaumesnil
  - Research Site, Beaumont-en-Véron
  - Research Site, Beauzelle
  - Research Site, Belfort
  - Research Site, Bellac
  - Research Site, Belleville-sur-Meuse
  - Research Site, Belz
  - Research Site, Bergholtz
  - Research Site, Bernin
  - Research Site, Beynes
  - Research Site, Bezons
  - Research Site, Bélâbre
  - Research Site, Bérat
  - Research Site, Bétaille
  - Research Site, Béthune
  - Research Site, Béville-le-Comte
  - Research Site, Béziers
  - Research Site, Biganos
  - Research Site, Bignan
  - Research Site, Billy-Montigny
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanquefort
  - Research Site, Blanzat
  - Research Site, Blénod-lès-Pont-à-Mousson
  - Research Site, Blois
  - Research Site, Bobigny
  - Research Site, Boën-sur-Lignon
  - Research Site, Bois de Nefles Saint Paul
  - Research Site, Bois-le-Roi
  - Research Site, Boiscommun
  - Research Site, Bompas
  - Research Site, Bondues
  - Research Site, Bonsecours
  - Research Site, Boos
  - Research Site, Boujan-sur-Libron
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourbriac
  - Research Site, Bourg de Joué-sur-Erdre
  - Research Site, Bourg-Achard
  - Research Site, Bourg-de-Péage
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourron-Marlotte
  - Research Site, Bourth
  - Research Site, Bousse
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Breuil-le-Sec
  - Research Site, Bréhal
  - Research Site, Briançon
  - Research Site, Brie
  - Research Site, Brienne-le-Château
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bruay-la-Buissière
  - Research Site, Cabannes
  - Research Site, Caen
  - Research Site, Callian
  - Research Site, Caluire-et-Cuire
  - Research Site, Camors
  - Research Site, Cannes La Bocca
  - Research Site, Canteleu
  - Research Site, Capbreton
  - Research Site, Carantec
  - Research Site, Carbon-Blanc
  - Research Site, Carhaix-Plouguer
  - Research Site, Carmaux
  - Research Site, Carnon-Plage
  - Research Site, Carquefou
  - Research Site, Carresse-Cassaber
  - Research Site, Carros
  - Research Site, Castets-en-Dorthe
  - Research Site, Castres
  - Research Site, Cauchy-à-la-Tour
  - Research Site, Caussade
  - Research Site, Cavaillon
  - Research Site, Celles-sur-Plaine
  - Research Site, Cernay
  - Research Site, Cérences
  - Research Site, Chaillevette
  - Research Site, Chalais
  - Research Site, Chalamont
  - Research Site, Chambéry
  - Research Site, Chambray-lès-Tours
  - Research Site, Champagne-sur-Oise
  - Research Site, Champagnole
  - Research Site, Champigné
  - Research Site, Champigny-sur-Marne
  - Research Site, Chanac
  - Research Site, Chapelle Saint Martin Plaine
  - Research Site, Charleville-Mézières
  - Research Site, Charvieu-Chavagneux
  - Research Site, Chassieu
  - Research Site, Chauvigny
  - Research Site, Chavanges
  - Research Site, Châbons
  - Research Site, Château-d'Olonne
  - Research Site, Château-Thierry
  - Research Site, Châteaubriant
  - Research Site, Châteaugay
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châtillon-Coligny
  - Research Site, Châtillon-Saint-Jean
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Châtillon-sur-Seine
  - Research Site, Chelles
  - Research Site, Chenôve
  - Research Site, Cherves-Richemont
  - Research Site, Choisey
  - Research Site, Ciboure
  - Research Site, Clairac
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Colombes
  - Research Site, Combrit
  - Research Site, Comines
  - Research Site, Commentry
  - Research Site, Concarneau
  - Research Site, Conty
  - Research Site, Corbehem
  - Research Site, Cordes-sur-Ciel
  - Research Site, Corseul
  - Research Site, Coudekerque-Branche
  - Research Site, Couhé
  - Research Site, Coulommiers
  - Research Site, Courcy
  - Research Site, Coursan
  - Research Site, Coussac-Bonneval
  - Research Site, Coye-la-Forêt
  - Research Site, Créteil
  - Research Site, Criquetot-l'Esneval
  - Research Site, Crolles
  - Research Site, Cugnaux
  - Research Site, Cuise-la-Motte
  - Research Site, Culoz
  - Research Site, Dambach-la-Ville
  - Research Site, Danjoutin
  - Research Site, Dessenheim
  - Research Site, Dieppe
  - Research Site, Dijon
  - Research Site, Domène
  - Research Site, Drancy
  - Research Site, Drap
  - Research Site, Dunkirk
  - Research Site, Ecques
  - Research Site, Einville-au-Jard
  - Research Site, Enghien-les-Bains
  - Research Site, Entre Deux
  - Research Site, Esquerdes
  - Research Site, Eu
  - Research Site, Eygalières
  - Research Site, Eyragues
  - Research Site, Épernon
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Feurs
  - Research Site, Firmi
  - Research Site, Firminy
  - Research Site, Fitilieu
  - Research Site, Fitz-James
  - Research Site, Flers
  - Research Site, Fleury-les-Aubrais
  - Research Site, Fleury-sur-Andelle
  - Research Site, Fléville-devant-Nancy
  - Research Site, Florange
  - Research Site, Folembray
  - Research Site, Fontaine
  - Research Site, Fos-sur-Mer
  - Research Site, Fougères
  - Research Site, Fouras
  - Research Site, Fourchambault
  - Research Site, Frontenas
  - Research Site, Frotey-lès-Vesoul
  - Research Site, Gaillon
  - Research Site, Gallardon
  - Research Site, Gardonne
  - Research Site, Garéoult
  - Research Site, Gauriac
  - Research Site, Gelles
  - Research Site, Gelos
  - Research Site, Gennes
  - Research Site, Gennevilliers
  - Research Site, Gignac-la-Nerthe
  - Research Site, Givors
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gonneville-la-Mallet
  - Research Site, Gorron
  - Research Site, Goudelin
  - Research Site, Gourdon
  - Research Site, Grand-Bois
  - Research Site, Grane
  - Research Site, Granville
  - Research Site, Graulhet
  - Research Site, Grignols
  - Research Site, Guenrouet
  - Research Site, Guéret
  - Research Site, Guignicourt
  - Research Site, Guise
  - Research Site, Guitalens-L'Albarède
  - Research Site, Hagondange
  - Research Site, Ham
  - Research Site, Hanvec
  - Research Site, Hénin-Beaumont
  - Research Site, Houilles
  - Research Site, Hulluch
  - Research Site, Hundling
  - Research Site, Inchy
  - Research Site, Isle
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivry-sur-Seine
  - Research Site, Jacou
  - Research Site, Jargeau
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jassans-Riottier
  - Research Site, Joncherey
  - Research Site, Jonquières-Saint-Vincent
  - Research Site, Jouy-le-Châtel
  - Research Site, Jugon-les-Lacs
  - Research Site, Jussey
  - Research Site, Knutange
  - Research Site, L Etang Sale
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Isle-Jourdain
  - Research Site, La Baule-Escoublac
  - Research Site, La Bâtie-Neuve
  - Research Site, La Bretagne
  - Research Site, La Broque
  - Research Site, La Cambe
  - Research Site, La Chapelle-des-Marais
  - Research Site, La Chapelle-en-Serval
  - Research Site, La Courneuve
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Fère
  - Research Site, La Forêt-sur-Sèvre
  - Research Site, La Fouillade
  - Research Site, La Francheville
  - Research Site, La Garde
  - Research Site, La Garenne-Colombes
  - Research Site, La Haye-Pesnel
  - Research Site, La Madeleine
  - Research Site, La Mothe-Saint-Héray
  - Research Site, La Motte-Servolex
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Talaudière
  - Research Site, La Teste-de-Buch
  - Research Site, La Tour-de-Salvagny
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, Labarthe-sur-Lèze
  - Research Site, Labenne
  - Research Site, Lagarde-Enval
  - Research Site, Lamagistère
  - Research Site, Lamalou-les-Bains
  - Research Site, Lançon-Provence
  - Research Site, Landerneau
  - Research Site, Landéan
  - Research Site, Landouge
  - Research Site, Lannion
  - Research Site, Lanouaille
  - Research Site, Laroquebrou
  - Research Site, Laudun-lArdoise
  - Research Site, Laval
  - Research Site, Lavelanet
  - Research Site, Le Barcarès
  - Research Site, Le Bois-dOingt
  - Research Site, Le Cailar
  - Research Site, Le Cannet
  - Research Site, Le Château-d’Oléron
  - Research Site, Le Grand-Lucé
  - Research Site, Le Grand-Quevilly
  - Research Site, Le Guillaume
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Langon
  - Research Site, Le Lavandou
  - Research Site, Le Luc
  - Research Site, Le Mée-sur-Seine
  - Research Site, Le Plessis-Bouchard
  - Research Site, Le Plessis-Robinson
  - Research Site, Le Pontet
  - Research Site, Le Port
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Rouret
  - Research Site, Le Teich
  - Research Site, Le Teil
  - Research Site, Le Tignet
  - Research Site, Le Trait
  - Research Site, Lectoure
  - Research Site, Leers
  - Research Site, Lembach
  - Research Site, Les Clayes-sous-Bois
  - Research Site, Les Forges
  - Research Site, Les Mureaux
  - Research Site, Les Paroches
  - Research Site, Les Sables-d'Olonne
  - Research Site, Leyme
  - Research Site, Lezoux
  - Research Site, Lédignan
  - Research Site, Lézardrieux
  - Research Site, Liffré
  - Research Site, Lignan-sur-Orb
  - Research Site, Ligny-en-Barrois
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Limogne-en-Quercy
  - Research Site, Livry-Gargan
  - Research Site, Loches
  - Research Site, Lognes
  - Research Site, Louverné
  - Research Site, Louvigné-du-Désert
  - Research Site, Ludon-Médoc
  - Research Site, Lunel
  - Research Site, Lunel-Viel
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Lussac-les-Châteaux
  - Research Site, Lyon
  - Research Site, Lys-lez-Lannoy
  - Research Site, Magland
  - Research Site, Mainvilliers
  - Research Site, Maisons-Alfort
  - Research Site, Maisons-Laffitte
  - Research Site, Malakoff
  - Research Site, Malemort-du-Comtat
  - Research Site, Malemort-sur-Corrèze
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Manduel
  - Research Site, Marange-Silvange
  - Research Site, Marciac
  - Research Site, Marckolsheim
  - Research Site, Marcq-en-Barœul
  - Research Site, Mareuil-sur-Lay-Dissais
  - Research Site, Marignane
  - Research Site, Marle
  - Research Site, Marlenheim
  - Research Site, Marly
  - Research Site, Marmande
  - Research Site, Marquion
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseille
  - Research Site, Martigues
  - Research Site, Martin-Église
  - Research Site, Mas-Grenier
  - Research Site, Masevaux
  - Research Site, Matha
  - Research Site, Mauguio
  - Research Site, Mauléon-Licharre
  - Research Site, Maurecourt
  - Research Site, Maxéville
  - Research Site, Mazan
  - Research Site, Mensignac
  - Research Site, Metz
  - Research Site, Meudon
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meursault
  - Research Site, Mezzavia
  - Research Site, Méjannes-lès-Alès
  - Research Site, Méounes-lès-Montrieux
  - Research Site, Mérignac
  - Research Site, Mézidon-Canon
  - Research Site, Mézilles
  - Research Site, Miramas
  - Research Site, Mirande
  - Research Site, Moncé-en-Belin
  - Research Site, Moncontour de Bretagne
  - Research Site, Monéteau
  - Research Site, Mons-en-Laonnois
  - Research Site, Montauban
  - Research Site, Montauroux
  - Research Site, Montbrison
  - Research Site, Montendre
  - Research Site, Montesson
  - Research Site, Monteux
  - Research Site, Montfavet
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montmagny
  - Research Site, Montmorillon
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montreuil-sur-Ille
  - Research Site, Montrevel-en-Bresse
  - Research Site, Montry
  - Research Site, Moreuil
  - Research Site, Morlaix
  - Research Site, Mortagne-du-Nord
  - Research Site, Morteau
  - Research Site, Mourioux-Vieilleville
  - Research Site, Moussy-le-Neuf
  - Research Site, Moutiers-les-Mauxfaits
  - Research Site, Mouvaux
  - Research Site, Mouy
  - Research Site, Moyaux
  - Research Site, Moyeuvre-Grande
  - Research Site, Mulhouse
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Neufchef
  - Research Site, Neuville-Saint-Rémy
  - Research Site, Nègrepelisse
  - Research Site, Néré
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-le-Phaye
  - Research Site, Nogent-le-Rotrou
  - Research Site, Noirmoutier-en-l'Île
  - Research Site, Noisy-le-Grand
  - Research Site, Nomain
  - Research Site, Nouâtre
  - Research Site, Noyelles-sous-Lens
  - Research Site, Noyen-sur-Sarthe
  - Research Site, Oberhausbergen
  - Research Site, Olby
  - Research Site, Orchies
  - Research Site, Orcines
  - Research Site, Origny Ste Benoite
  - Research Site, Orléans
  - Research Site, Orly
  - Research Site, Ormes
  - Research Site, Orthez
  - Research Site, Orvault
  - Research Site, Ouroux-sur-Saône
  - Research Site, Oyonnax
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paimpol
  - Research Site, Pantin
  - Research Site, Parcey
  - Research Site, Paris
  - Research Site, Parthenay
  - Research Site, Pau
  - Research Site, Peaugres
  - Research Site, Pernes-les-Fontaines
  - Research Site, Perpignan
  - Research Site, Perros-Guirec
  - Research Site, Petite-Synthe
  - Research Site, Pérenchies
  - Research Site, Pfaffenhoffen
  - Research Site, Pisany
  - Research Site, Plaisance-du-Touch
  - Research Site, Pleaux
  - Research Site, Plélan-le-Grand
  - Research Site, Plérin
  - Research Site, Ploemeur
  - Research Site, Ploeren
  - Research Site, Pocé-sur-Cisse
  - Research Site, Pont-de-Buis-lès-Quimerch
  - Research Site, Pont-Évêque
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pontailler-sur-Saône
  - Research Site, Pontault-Combault
  - Research Site, Pontivy
  - Research Site, Pornic
  - Research Site, Port-de-Bouc
  - Research Site, Port-La Nouvelle
  - Research Site, Potigny
  - Research Site, Pouilley-les-Vignes
  - Research Site, Pouilly-en-Auxois
  - Research Site, Poussan
  - Research Site, Privas
  - Research Site, Provins
  - Research Site, Puteaux
  - Research Site, Puygouzon
  - Research Site, Quarouble
  - Research Site, Questembert
  - Research Site, Quiberon
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quincy-Voisins
  - Research Site, Rabastens-de-Bigorre
  - Research Site, Rambervillers
  - Research Site, Rebais
  - Research Site, Reims
  - Research Site, Réding
  - Research Site, Richardménil
  - Research Site, Rieupeyroux
  - Research Site, Rieux
  - Research Site, Rilhac-Rancon
  - Research Site, Rivery
  - Research Site, Roanne
  - Research Site, Robion
  - Research Site, Rognes
  - Research Site, Rohrwiller
  - Research Site, Roissy-en-France
  - Research Site, Romagnat
  - Research Site, Romainville
  - Research Site, Rombas
  - Research Site, Romilly-sur-Seine
  - Research Site, Romorantin-Lanthenay
  - Research Site, Roncey
  - Research Site, Roncq
  - Research Site, Rosières
  - Research Site, Rosières-en-Santerre
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rouillac
  - Research Site, Routot
  - Research Site, Royan
  - Research Site, Sains-du-Nord
  - Research Site, Saint Georges Baillargeaux
  - Research Site, Saint Gilles Les Bains
  - Research Site, Saint Gilles Les Hauts
  - Research Site, Saint Maximin La Ste Baume
  - Research Site, Saint-Affrique
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubert
  - Research Site, Saint-Aubin-des-Châteaux
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Barthélémy
  - Research Site, Saint-Beauzire
  - Research Site, Saint-Benoît
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Claude-de-Diray
  - Research Site, Saint-Clément
  - Research Site, Saint-Cyprien
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-lès-Bourg
  - Research Site, Saint-Erme-Outre-et-Ramecourt
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-lès-Remiremont
  - Research Site, Saint-Genest-Malifaux
  - Research Site, Saint-Georges-des-Groseillers
  - Research Site, Saint-Germain-les-Belles
  - Research Site, Saint-Guénolé
  - Research Site, Saint-Herblain
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-du-Gard
  - Research Site, Saint-Jeannet
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Lambert-la-Potherie
  - Research Site, Saint-Laurent-Blangy
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Leu
  - Research Site, Saint-Léon-sur-l'Isle
  - Research Site, Saint-Mamert-du-Gard
  - Research Site, Saint-Marcel-lès-Valence
  - Research Site, Saint-Marcellin
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Max
  - Research Site, Saint-Médard-de-Guizières
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Pierre-de-Chandieu
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-en-Val
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Saëns
  - Research Site, Saint-Savinien
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Sylvain
  - Research Site, Saint-Yorre
  - Research Site, Saintes
  - Research Site, Salbris
  - Research Site, Salernes
  - Research Site, Salomé
  - Research Site, Salornay-sur-Guye
  - Research Site, Samer
  - Research Site, Sarreguemines
  - Research Site, Sarry
  - Research Site, Sars-Poteries
  - Research Site, Saulnot
  - Research Site, Sault-lès-Rethel
  - Research Site, Sauveterre-de-Rouergue
  - Research Site, Saverdun
  - Research Site, Savigny-le-Temple
  - Research Site, Savonnières
  - Research Site, Schiltigheim
  - Research Site, Schirrhein
  - Research Site, Segonzac
  - Research Site, Segré
  - Research Site, Sens
  - Research Site, Sens-de-Bretagne
  - Research Site, Seyssinet-Pariset
  - Research Site, Sète
  - Research Site, Sérifontaine
  - Research Site, Sérignan
  - Research Site, Simiane-Collongue
  - Research Site, Sissonne
  - Research Site, Six-Fours-les-Plages
  - Research Site, Socx
  - Research Site, Soissons
  - Research Site, Soisy-sous-Montmorency
  - Research Site, Solliès-Pont
  - Research Site, Solre-le-Château
  - Research Site, Sorcy-Saint-Martin
  - Research Site, St-Malo
  - Research Site, Stains
  - Research Site, Ste Anne
  - Research Site, Ste Clotilde
  - Research Site, Ste Fereole
  - Research Site, Ste Fortunade
  - Research Site, Ste Mere Eglise
  - Research Site, Ste Severe Sur Indre
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Tarbes
  - Research Site, Tence
  - Research Site, Terre Sainte
  - Research Site, Thann
  - Research Site, Thionville
  - Research Site, Thiviers
  - Research Site, Thouars
  - Research Site, Thun-Saint-Amand
  - Research Site, Tilly-sur-Seulles
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Traînel
  - Research Site, Traînou
  - Research Site, Tréguier
  - Research Site, Trévières
  - Research Site, Trith-Saint-Léger
  - Research Site, Troissereux
  - Research Site, Turretot
  - Research Site, Uckange
  - Research Site, Uxem
  - Research Site, Uzès
  - Research Site, Vailly-sur-Aisne
  - Research Site, Valence-d'Albigeois
  - Research Site, Valff
  - Research Site, Valras-Plage
  - Research Site, Vals-les-Bains
  - Research Site, Vaulx-en-Velin
  - Research Site, Veigné
  - Research Site, Velleron
  - Research Site, Venarey-les-Laumes
  - Research Site, Vendeuil
  - Research Site, Vendôme
  - Research Site, Verfeil
  - Research Site, Vernouillet
  - Research Site, Verquières
  - Research Site, Vertus
  - Research Site, Vervins
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vif
  - Research Site, Vigneux-sur-Seine
  - Research Site, Vihiers
  - Research Site, Ville-di-Pietrabugno
  - Research Site, Villefontaine
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranque
  - Research Site, Villejuif
  - Research Site, Villemeux-sur-Eure
  - Research Site, Villemomble
  - Research Site, Villeneuve-Tolosane
  - Research Site, Villepreux
  - Research Site, Villers-Bocage
  - Research Site, Villers-Bretonneux
  - Research Site, Villette-d'Anthon
  - Research Site, Villeurbanne
  - Research Site, Villiers-sur-Marne
  - Research Site, Vinay
  - Research Site, Vincennes
  - Research Site, Vitrolles
  - Research Site, Vitteaux
  - Research Site, Vivy
  - Research Site, Voisins-le-Bretonneux
  - Research Site, Voujeaucourt
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Wignehies
  - Research Site, Wittelsheim
  - Research Site, Yerville